CLINICAL TRIAL: NCT00746902
Title: Study of the Relationships Between Refractory Hypertension, Overweight/Obesity and Sleep Apnea Syndrome
Acronym: RHOOSAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation de Recherche sur l'Hypertension Artérielle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0803; 2008-A00292-53 (Registry Identifier: ID RCB)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Refractory Hypertension
Keywords: Refractory hypertension; Obstructive sleep apnea syndrome; Obesity; Leptinemia; RHOOSAS study
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Arm 1: Active CPAP, a nasal continuous positive airway pressure
  Interventions: Device: nCPAP
- 2 (Sham Comparator): Arm 2 : Sham CPAP :Placebo/CPAP
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: nCPAP — Active nCPAP

SUMMARY:
The purpose of the study is to investigate the links between blood pressure (BP), overweight or obesity, and sleep apnea syndrome (SAS), by studying a large cohort of subjects suffering from refractory hypertension.

Primary objective

* To compare plasmatic leptin levels in patients suffering from refractory hypertension depending on whether or not they experience SAS.

Secondary objectives

* To ascertain what determines the difference in plasmatic leptin concentrations in patients suffering from refractory hypertension depending on whether or not they experience SAS.
* To characterise BP readings (from clinical and ambulatory (ABPM) measurements) in patients suffering from refractory hypertension depending on whether or not they experience SAS.
* To characterise metabolic parameters (lipids, glycaemia, adiponectin) and sympathetic nervous system effectors (adrenaline, noradrenaline and metanephrines) in patients suffering from refractory hypertension depending on whether or not they experience SAS.
* To characterise BP readings, metabolic parameters and sympathetic nervous system effectors in patients suffering from refractory hypertension according to the severity of the SAS (in those who experience this problem).
* To study, in patients with both SAS and refractory hypertension, the impact of nasal continuous positive airway pressure (CPAP) treatment on BP readings, metabolic parameters and sympathetic nervous system effectors, by comparing those who are compliant with the CPAP regimen with those who are non-compliant.

DETAILED DESCRIPTION:
A number of factors predispose subjects to both hypertension and SAS, including overweight/obesity and hyperinsulinism. The pathogenesis of concomitant overweight/obesity and hypertension is multifactorial. There is an independent relationship between the degree of insulin resistance and the severity of SAS. A number of studies have suggested that hormones secreted by adipose tissue are involved in the pathogenesis of both hypertension and SAS, and overweight/obesity has been shown to be associated with elevated leptin levels coupled with reduced adiponectin levels.

Leptin is produced in adipose tissue and its levels rise with overweight/obesity due to peripheral resistance to its action. A number of studies have detected high leptinemia in both hypertensives and people suffering from SAS. Leptin may activate the sympathetic nervous system and promote SAS-related hypertension.

Adiponectin which is also produced in adipose tissue has beneficial activities, notably on atherogenesis. A relationship between hypertension and adiponectin has yet to be demonstrated.

Unlike leptin, adiponectin levels do not seem to be elevated in patients with SAS.

In terms of treatment, a number of studies have shown that CPAP has a positive effect on BP readings. Although this effect is modest, it is greater in subjects with SAS and rises with the severity of this condition. The effects of CPAP on plasmatic leptin and adiponectin levels are as yet unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, of between 18 and 70
* Suffering from refractory hypertension as defined by persistent clinical hypertension (> 140/90 mm Hg according to two different readings 24 hours apart) despite at least three classes of antihypertensive drugs (including a thiazide diuretic) at appropriate doses.
* Recruited in the Cardiology Departments of the University Hospitals in Grenoble, Toulouse, Marseille and Poitiers, and in the Mozart Clinic in Paris.
* Outpatients
* Patients who have signed the consent form
* Patients affiliated to or beneficiary of the social security system

Exclusion Criteria:

* Failure to fulfil the inclusion criteria
* Treated SAS, whatever the form of the treatment
* Disease which might affect BP regulation, including Parkinson's disease, kidney or heart transplantation, dysautonomia, severe heart failure
* Atrial fibrillation or regular extrasystole (> 10/minute)
* Night- or shift-work
* Pregnant and breast-feeding women
* Patients under legal guardianship
* Incarcerated patients or adults protected by the law
* Hospitalised patients
* Ongoing participation in another clinical research study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
leptinemia | inclusion visit, visit month 3, visit month 6 or 9

SECONDARY OUTCOMES:
BP readings (clinical and ABPM), metabolic parameters (lipids, glycaemia, adiponectin) and sympathetic nervous system effectors (adrenaline, noradrenaline and metanephrines). | inclusion visit, visit month 3, visit month 6 or 9

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe BAGUET, Professor, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Derived] Joyeux-Faure M, Baguet JP, Barone-Rochette G, Faure P, Sosner P, Mounier-Vehier C, Levy P, Tamisier R, Pepin JL. Continuous Positive Airway Pressure Reduces Night-Time Blood Pressure and Heart Rate in Patients With Obstructive Sleep Apnea and Resistant Hypertension: The RHOOSAS Randomized Controlled Trial. Front Neurol. 2018 May 8;9:318. doi: 10.3389/fneur.2018.00318. eCollection 2018. PMID 29867728